CLINICAL TRIAL: NCT02474485
Title: Absorb Bioresorbable Scaffold vs. Drug Coated Balloon for Treatment Of In-Stent-Restenosis
Brief Title: Absorb BVS vs. Drug Coated Balloon for Treatment Of ISR
Acronym: AbsorbISR
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Information of other studies with Abseb bioresorbable scaffolds showed a higher thrombotic risk than before, the risk for the Patients is estimated too high
Sponsor: SIS Medical AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AbsorbISR
Record Dates: First submitted 2015-06-11; First posted 2015-06-17 (Estimated); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Coronary Artery Disease; Coronary Restenosis
Keywords: bioresorbable vascular scaffold; Absorb; drug eluting balloon; percutaneous coronary intervention
MeSH Terms: conditions — Coronary Artery Disease; Coronary Restenosis | interventions — Watchful Waiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BVS - Absorb (Active Comparator): BVS - Absorb scaffold group will be treated by implantation of drug eluting bioresorbable vascular scaffold (Absorb®). In this arm following interventions will be performed:
  * BVS Absorb implantation. For in stent restenosis treatment during index procedure.
  * OCT visualization.During index procedure and at 9 month follow-up.
  * Control coronary angiography. Control angiography will be performed at 9 month follow-up.
  * Clinical observation. Clinical observation will be performed at 9, 12 and 60 month follow-up.
  Interventions: Device: BVS Absorb implantation.; Procedure: Control coronary angiography.; Procedure: OCT visualization.; Other: Clinical observation.
- DEB - Sequent Please (Active Comparator): In DEB - Sequent Please Group, dilatation of drug eluting balloon Sequent Please ® will be used for treatment of the narrowed part of the artery. In this arm following interventions will be performed:
  * DEB Sequent Please inflation. For in stent restenosis treatment during index procedure.
  * OCT visualization.During index procedure and at 9 month follow-up.
  * Control coronary angiography. Control angiography will be performed at 9 month follow-up.
  * Clinical observation. Clinical observation will be performed at 9, 12 and 60 month follow-up.
  Interventions: Device: DEB Sequent Please inflation.; Procedure: Control coronary angiography.; Procedure: OCT visualization.; Other: Clinical observation.

INTERVENTIONS:
Device: BVS Absorb implantation. — Absorb bioresorbable vascular scaffold will be implanted to treat in stent restenosis in target vessel.
  Arms: BVS - Absorb
Device: DEB Sequent Please inflation. — Inflation of drug eluting balloon Sequent Please will be performed to treat in stent restenosis in target vessel.
  Arms: DEB - Sequent Please
Procedure: Control coronary angiography. — Control coronary angiography will be performed at 9 month follow-up.
Procedure: OCT visualization. — OCT visualization will be performed during index procedure and at 9 month follow-up.
Other: Clinical observation. — Patients will be informed that Investigator will contact them at 12, 24 and 60 months after the procedure. Investigator will collect information regarding clinical status of Patients, cardiac medications and any adverse events that occurred since the last follow-up.

SUMMARY:
AbsorbISR is a randomized, controlled trial, single center, prospective, not blinded to evaluate two strategies of in stent restenosis treatment: Implantation of drug eluting bioresorbable stent scaffold Absorb® vs. balloon angioplasty with drug eluting balloon Sequent Please®.

DETAILED DESCRIPTION:
This is randomized-controlled trial of Absorb® Bioresorbable Vascular Scaffold (BVS) vs. Sequent Please® drug coated balloon in an all-comers population with in-stent-restenosis (ISR). The patients will be randomized in a 1:1 fashion and the investigators intend to include 150 patients.

All patients presenting with ISR and requiring percutaneous coronary intervention will be eligible to be included in this study. This will include patients with stable angina and those presenting with acute coronary syndrome (ACS).

The primary objective of this study is to demonstrate superiority of the Absorb® bioresorbable scaffold compared to the Sequent Please® Drug Coated Balloon when treating patients with In-Stent-Restenosis regards to primary endpoint - angiographic late lumen loss at 9 month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 18 years or above.
* Diagnosed with ISR requiring percutaneous coronary intervention: visual diameter stenosis > 70 % and/or Fractional Flow Reserve < 0.81 and/or non-invasive testing demonstrating ischemia. This real-life population with in-stent restenosis beside typical stable patients with ISR includes ACS patients with thrombus containing lesions, patients with multivessel disease, patients with ISR in non-infarct related artery, with ISR in bare metal stent (BMS), drug eluting stent (DES) or bioresorbable vascular scaffold (BVS), ISR in lesion previously treated by plain old balloon angioplasty (POBA), drug eluting balloon (DEB) or additional stent implantation.
* Double anti-platelet therapy for the duration of at least 12 months is considered possible at the time of intervention

Exclusion Criteria:

* The participant may not enter the study if the interventionist has doubts that he is not able to deliver and implant the Absorb scaffold (e.g. highly calcified lesions).
* Patients who have any contraindications for using DEB (SeQent Please) or BVS (Absorb) specified in instructions for use are not able to participate in this study.
* Women with childbearing potential must have a negative result of pregnancy test and they must use an effective contraception method for at least 12 months after study procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2015-03; Primary Completion 2018-05 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Angiographic late lumen loss at 9 month follow-up. | At 9 month follow up.
  Angiographic late lumen loss will be compared between both study groups.

SECONDARY OUTCOMES:
Incidence of periprocedural complications: unplanned use of GP IIb/IIIa inhibitors. | Participants will be followed for the duration of index procedure, an expected average of 1 hour.
Incidence of periprocedural complications: vessel rupture. | Participants will be followed for the duration of index procedure, an expected average of 1 hour.
Incidence of periprocedural complications: side branch occlusion. | Participants will be followed for the duration of index procedure, an expected average of 1 hour.
Incidence of periprocedural complications: peri-procedural myocardial infarction. | Participants will be followed for the duration of index procedure, an expected average of 1 hour.
Comparison of minimal luminal diameter between both groups and in specific populations (patients with acute coronary syndromes, patients with diabetes, patients with long lesions (> 25 mm)). | Participants will be followed for the duration of index procedure, an expected average of 1 hour.
Comparison of diameter stenosis between both groups and in specific populations (patients with acute coronary syndromes, patients with diabetes, patients with long lesions (> 25 mm)). | Participants will be followed for the duration of index procedure, an expected average of 1 hour.
Comparison of rate of restenosis between both groups and in specific populations (patients with acute coronary syndromes, patients with diabetes, patients with long lesions (> 25 mm)). | Participants will be followed for the duration of index procedure, an expected average of 1 hour.
Incidence of in-stent-restenosis in long-term observation. | During 60 month follow-up.
Incidence of target lesion failure in long-term observation. | During 60 month follow-up.
Incidence of target vessel revascularisation in long-term observation. | During 60 month follow-up.
Incidence of stent thrombosis in long-term observation. | During 60 month follow-up.
Occurence of stent thrombosis (defined as early, late and very late probable or definite according to ARC definition). | During 60 month follow-up.
Cardiac and non-cardiac death in both groups. | During 60 month follow-up.
Assessment of possibility vessel measurement and stent diameter/length choice based on these measurement in optical coherence tomography (OCT). | Participants will be followed for the duration of index procedure, an expected average of 1 hour.
Result of index procedure assessment in OCT post procedure (lumen/stent area, struts assessment, dissections, stent expansion). | Participants will be followed for the duration of index procedure, an expected average of 1 hour.
OCT assessment of long-term study results (lumen/stent area, struts assessment, neointimal volume, lumen volume). | At 9 month follow-up.
Lumen volume change between index and 9 month follow-up OCT. | OCT parameters change will be assessed between index hospitalization and 9 month follow-up.
Minimal lumen area change between index and 9 month follow-up OCT. | OCT parameters change will be assessed between index hospitalization and 9 month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Florim Cuculi, Prof. dr, Principal Investigator
Locations (1):
- Luzernen Kantonsspital, Spitalstrasse 16, Lucerne, Switzerland